CLINICAL TRIAL: NCT03361423
Title: A Randomized, Double Blinded, Sham Controlled Clinical Study to Evaluate the Safety and Efficacy of the Nerivio Migra 1, a Neuromodulation Device, for the Acute Treatment of Migraine
Brief Title: Evaluation of a Novel Device for Treatment of Migraine Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranica (Industry)
Collaborators: Rambam Health Care Campus (Other); Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCH003
Record Dates: First submitted 2017-11-18; First posted 2017-12-04 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2019-02

CONDITIONS: Migraine Without Aura; Migraine With Aura
MeSH Terms: conditions — Migraine without Aura; Migraine with Aura

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double blinded, sham controlled study
Who Masked: Participant, Investigator
Masking Description: For sham control, electrical pulses of similar width and intensity, but much lower frequency compared to the active device will be administered. This sham program produces pulses that are perceivable by the user, thus maintaining the blinding, but on the other hand do not have therapeutic qualities.
  The devices will be delivered with an identifying number, without exposing to the investigator or participant if it is an active or a pacebo/sham device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- treatment of migraine with active device (Active Comparator): Treatment of acute migraine with an active form of Nerivio migra-1 device
  Interventions: Device: Nerivio Migra-1 active device
- treatment of migraine with sham device (Sham Comparator): Treatment of acute migraine with a sham form of the Nerivio Migra-1 device
  Interventions: Device: Nerivio Migra-1 Sham device

INTERVENTIONS:
Device: Nerivio Migra-1 active device — The device is placed on the subject upper arm. when activated, stimulus is applied to influence the subject's perception of a painful stimulus, delivered (or originating) at a different location. Based on diffused noxious inhibitory control mechanism, sometimes referred to as "pain inhibits pain" principle, conditioned pain modulation evokes an endogenous analgesic mechanism. The modulatory effect is over the whole body, and can be induced anywhere in the body. This approach allows applying the conditioning stimuli away from the painful site.
  Arms: treatment of migraine with active device
Device: Nerivio Migra-1 Sham device — The device is placed on the subject upper arm. when activated, the stimulus is applied is not sufficient to influence the subject's perception of a painful stimulus.
  Arms: treatment of migraine with sham device

SUMMARY:
Migraine is a common neurologic with attacks of headache and associated symptoms such as nausea, vomiting, phono and photophobia. Migraine can lead to substantial functional impairment.

Recent evidence suggests that electro stimulation is effective in providing relief for chronic headaches including migraine. It is tolerable by patients and associated with no adverse effects.

The device utilizes electro stimulation to achieve conditioned pain modulation (CPM). CPM an stimulate endogenous analgesic mechanism. The modulatory effect is over the whole body, and can be induced anywhere.

This is a prospective, randomized, double-blind, sham controlled multi-center trial. Ratio between treatment and control groups will be 1:1, stratified by center and use of preventive medications.

The study objectives is to demonstrate the safety and effectiveness of the Nerivio Migra electro stimulation device for the reduction of migraine headache during an attack of migraine with or without aura.

The study is intended for subject with 2-8 migraine episodes per month. patients will receive the device, either an active or a placebo type, and will be asked to use the device at home or in any location that they will be when the migraine starts.

The study hypothesis is that electro stimulation delivered transcutaneously to the peripheral nervous system at onset of a migraine attack significantly reduce headache pain demonstrated by a significant difference between proportions of responders to the active treatment stimulation in comparison to proportion of responders that will use a placebo device.

DETAILED DESCRIPTION:
Nerivio Migra is intended for the acute treatment of migraine with or without aura in patients 18 years of age or older. It is self-applied to the upper arm. Treatments are self-administered by the user at the onset of a migraine attack. The device delivers extra cephalic transcutaneous electrical stimulation below the pain threshold to the skin of the upper arm at the onset of a migraine attack. Nerivio Migra is operated via a mobile application.

This is a prospective, randomized, double-blind, sham controlled multi-center clinical trial to test the ability of the Nerivio Migra neuromodulation device to relieve the patient's migraine pain during a migraine attack. The study will enroll up to 270 patients diagnosed with migraine with or without aura, per the inclusion and exclusion criteria. These patients will be individually and randomly assigned to either treatment group or control group. For sham control, electrical pulses of similar width and intensity, but much lower frequency compared to the active device will be administered. This sham program produces pulses that are perceivable by the user, thus maintaining the blinding, but on the other hand do not have therapeutic qualities, based on existing knowledge of parameters range of electro stimulation treatments.

1. st visit - screening, enrollment and training on the application in diary mode Following successful screening, enrollment interview and signing of informed consent, participants will be provided with the Nerivio Migra application (either installed on their own smartphone, or on a smartphone provided by the study coordinator). The participants will be trained how to operate the application and report their migraine attacks in the patient diary mode, which is part of the application. The site personnel will be required to approve the training session in the CRF.

   Stage 1 - Roll in phase The Roll-in is a period of 15 - 30 days in which at least two (2) and no more of eight (8) migraine attacks has been occurred. During this period, baseline information including mean frequency and severity of migraine attacks, occurrence of other headaches, presence of ICHD-3 diagnostic criteria for migraine with or without aura and use of preventive and rescue medications will be recorded.
2. nd visit Following the Roll-in phase, the participants will arrive to the clinic and their compliance to the study procedures and eligibility to continue to the next phase will assessed.

Participants that will be eligible to continue to the treatment phase will undergo the following:

1. Participant will be randomized into one of the two study group (Active or Sham device) Investigational devices will be programmed in active or sham mode with a 1:1 ratio, in order to achieve the desired ratio between active and control groups sizes, stratified with by use of preventive medications.
2. Participant will be trained on the device, the application (in diary and treatment modes), the treatment procedures and the key elements critical for the success of the study:

   * Apply the Nerivio Migra as soon as possible following the onset of the migraine symptoms and NO LATER than 60 min from onset
   * Refrain from taking any rescue medication 2 hours following the start of treatment.
   * Perform the treatment for a period of at least 30 minutes (recommended treatment time is 45 minutes).

Stage 2 - Parallel arms, double- blind treatment phase. Participants will be instructed to activate the device at onset of a qualifying migraine attack and manually adjust stimulation intensity to a level within the pre-defined range, where it is well perceived but not painful. A qualifying migraine attack shall be preceded by at least 48 hours of freedom from migraine. Patients will be requested to refrain from use of rescue medications prior to and during the first two hours after treatment with the device, and if they cannot comply with this, record their use of rescue medications (migraine specific drugs or other medications or therapies that may be used to treat pain, from a pre-specified list) in the mobile application.

Via the smartphone application, each participant will be asked to rate his/her migraine pain level three times using Pain Grades Scale (0 - no pain, 1- mild pain, 2- moderate pain, 3 - severe pain): (1) upon starting the treatment, (2) two hours after start of treatment, (3) 48 hours after start of attack. At the start of each treatment, participants will be also asked to provide time elapsed from start of migraine symptoms to start of the treatment. Participants will be also asked to provide feedback regarding their use of medication (migraine specific drugs or other medications or therapies that may be used to treat pain, from a pre-specified list), presence of nausea, photophobia, phonophobia or allodynia, and treatment perception. After providing feedback at two hours after start of treatment and in case of pain recurrence, participants will be allowed to re-treat the attack using Nerivio Migra device.

Adverse events will be reported.

Stage 3 (optional, by subject request only) - Open label extended treatment:

Following the completion of double-blind stage of the study, all subjects will be offered a 2-month open label period using the active device.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18-75 years old.
2. Subjects meet the ICHD-3 diagnostic criteria for migraine with or without aura
3. Subjects report 2-8 migraine attacks per month.
4. Stable migraine preventive medications in the last two months prior to recruitment (No change in usage or dosage).
5. Subjects must be able and willing to comply with the protocol
6. Subjects must be able and willing to provide written informed consent

Exclusion Criteria:

1. Subject has other significant pain, medical or psychologic problems that in the opinion of the investigator may confound the study assessments
2. Subject has an implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagus nerve neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator).
3. Subject has known uncontrolled epilepsy.
4. Any use of Cannabis including medical use.
5. Subject has >10 headache days per month.
6. Subject has undergone nerve block (occipital or other) in the head or neck within the last 2 weeks.
7. Subject is participating in any other clinical study.
8. The subject does not have the basic cognitive and motor skills needed to operate a smartphone.
9. Pregnant, or trying to get pregnant
10. Subject is experiencing a menstrually related migraine
11. Received OnabotulinumtoxinA or any botulinum toxin injections for migraine within the previous month
12. Received parenteral infusions for migraine within the previous 2 weeks.
13. Subject participated in a previous study with the Nerivio Migra 1 device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, Prof, Study Director — Rambam Medical Center, Israel; Moris Levin, MD, Study Chair — University California Sun Francisco, USA
Locations (12):
- United States (7):
  - Hartford Headache Center, Hartford, Connecticut
  - Clinvest Research, Springfield, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Clinical Reseach Consortium, Las Vegas, Nevada
  - Northwell Health, Inc, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Israel (5):
  - Rambam Medical Center, Haifa
  - wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Belinson Medical Center, Petah Tikva
  - Souraskyr Medical center - Ichilov, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rapoport AM, Bonner JH, Lin T, Harris D, Gruper Y, Ironi A, Cowan RP. Remote electrical neuromodulation (REN) in the acute treatment of migraine: a comparison with usual care and acute migraine medications. J Headache Pain. 2019 Jul 22;20(1):83. doi: 10.1186/s10194-019-1033-9. PMID 31331265
- [Derived] Yarnitsky D, Dodick DW, Grosberg BM, Burstein R, Ironi A, Harris D, Lin T, Silberstein SD. Remote Electrical Neuromodulation (REN) Relieves Acute Migraine: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial. Headache. 2019 Sep;59(8):1240-1252. doi: 10.1111/head.13551. Epub 2019 May 9. PMID 31074005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: a 4 weeks "run-in" phase. during this phase, participants recorded their migraine attacks and complete a migraine diary at T=0,2 and 48 hours for each migraine attack.
  Participant who had 2-8 attacks and completed at least 66% of their migraine diary were eligible to continue to the treatment phase
Period: Overall Study
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Started | 126 | 126
Completed | 99 | 103
Not Completed | 27 | 23
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Did not treat | 19 | 18
Not completed — Started >60 minutes from migraine onset | 0 | 1
Not completed — Missing data | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device | Total
Number analyzed (Participants) | 126 | 126 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.25) | 41.6 (11.81) | 42.7 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 102 | 203
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 10 | 8 | 18
  White | 109 | 112 | 221
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90 | 85 | 175
  Israel | 36 | 41 | 77
Average number of migraines attacks per month [Mean (Standard Deviation); unit: Attacks per month] | 5.2 (1.95) | 5.3 (1.90) | 5.3 (1.92)
Average number of migraine days per month [Mean (Standard Deviation); unit: Days per month] | 6.6 (2.43) | 6.6 (2.41) | 6.6 (2.40)
Use of preventive medication [Count of Participants; unit: Participants] | 36 | 46 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reduction of Migraine Headache at 2 Hours Post Treatment
Description: The percentage of patients reporting reduction in their pain level 2 hours post-treatment without rescue medications from severe or moderate to mild or no pain, or from mild to no pain, in their first treated migraine attack (excluding the "run-in test" treatment).
Time Frame: 2 hours post migraine onset
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 99 | 103
Participants | 66 | 40

2. Secondary Outcome: Percentage of Participants With Reduction of Most Bothersome Migraine-associated Symptom (MBS) Relief at 2 Hours Post Treatment
Description: The percentage of patients reporting, 2 hours post-treatment, freedom from their most bothersome migraine-associated symptom (MBS) other than a headache, in their first treated migraine attack (excluding the "run-in test" treatment). MBS may be nausea, photophobia, phonophobia or allodynia - as defined by each subject at the beginning of the treatment
Time Frame: 2 hours post migraine onset
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 95 | 99
Participants | 44 | 22

3. Secondary Outcome: Percentage of Participants With Reduced Migraine Headache AND MBS Relief at 2 Hours Post Treatment
Description: The percentage of patients reporting, 2 hours post treatment response to both the primary and the first secondary endpoints
Time Frame: 2 hours post migraine onset
Population: 4 participants in the active group and 4 participants in the sham group did not report their MBS level at the beginning of the treatment or at 2 hours post treatment. Thus, the active and sham groups included 95 and 99 participants, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 95 | 99
Participants | 38 | 15

4. Secondary Outcome: Percentage of Participants With Pain Disappearance at 2 Hours Post Treatment
Description: The percentage of subjects reporting freedom from migraine pain at 2 hours post-treatment without medications in their first treated migraine attack
Time Frame: 2 hours post migraine onset
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 99 | 103
Participants | 37 | 19

5. Other Pre Specified Outcome: Number of Adverse Events Related or Unrelated to the Study Device
Description: The number of Adverse events related to the study device. Safety analyses were performed on all participants from the ITT population (126 participants in each group).
Time Frame: up to 14 weeks
Measure: Number; unit: Adverse event
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 126 | 126
Adverse event | 14 | 9

6. Other Pre Specified Outcome: Within-patient Consistency - Percentage of Participants With Reduction in Headache Pain in at Least 50% of Their Treatments
Description: The repeatability of migraine headache reduction, as described in the primary endpoint definition, in subsequent treated attacks. Thus, this endpoint measures the % of patient responding to the primary endpoint in at least 50% of their treated attacks (excluding the run-in attack
Time Frame: up to 6 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 99 | 103
percentage of participants | 51.3 [42.8 to 61.4] | 38.1 [31.2 to 46.6]

7. Other Pre Specified Outcome: Percentage of Participants With Sustained Pain-free 48 Hours With Single Use of the Device
Description: The proportion (%) of subjects reporting pain-free at 2 hours, and no return of any pain or use of rescue/acute medication, or reuse of device between 2 hours and 48 hours, in their first treated migraine attack
Time Frame: 48 hours post treatment
Population: 12 participants in the active group and 14 participants in the sham group did not report their pain level at 24h post treatment for the "Test" treatment. Thus, the active and sham groups included 87and 89 participants, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 87 | 89
Participants | 18 | 6

8. Other Pre Specified Outcome: Percentage of Participants With Sustained Headache Reduction for 48 Hours With Single Use of the Device
Description: The proportion (%) of subjects reporting treatment response 2 hours post-treatment without rescue medications, and no return to baseline level of pain at time of treatment, or use of rescue/acute medication, or reuse of device between 2 hours and 48 hours, in their first treated migraine attack
Time Frame: 48 hours post treatment
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
Number analyzed (Participants) | 87 | 89
Participants | 32 | 14

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Description: The Nerivio device is a neurostimulator and it is externally applied over the body. The Nerivio is accepted as a non-significant risk (NSR) device. In addition, as the exclusion criteria for the study leave out participant with electrical implant, congenital heart failure or epilepsy, the number of high risk participants is zero.
Arm/Group | Treatment of Migraine With Active Device | Treatment of Migraine With Sham Device
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/126
Other Adverse Events (participants affected / at risk) | 14/126 | 9/126
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment of Migraine With Active Device (N=126) | Treatment of Migraine With Sham Device (N=126)
Sensation of warmth (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Numbness of the arm (Nervous system disorders) | 2 (2) | 0 (0)
Pain in the arm (Nervous system disorders) | 2 (2) | 0 (0)
Redness of the skin at the treatment area (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Neck and shoulder pain (Product Issues) | 0 (0) | 2 (2)
Tingling (Product Issues) | 0 (0) | 3 (3)
Muscle spasm (Nervous system disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03361423/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03361423/ICF_001.pdf